CLINICAL TRIAL: NCT04135885
Title: Effect of Preoperative Folic Acid Intervention on Postoperative Recovery Period in Children With Head and Neck and Maxillofacial Surgery
Brief Title: Folic Acid Intervention During Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SH9H-2019-T122
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Adverse Effect of Other General Anesthetics
Keywords: Folic Acid; Placebo
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: patients took 7 days of folic acid tablets before surgery (0.3mg/d for children aged 1-3, 0.4mg/d for children aged 4~5 years, dissolved in 20ml brown sugar water.)
  Interventions: Drug: Folic Acid
- Placebo group (Experimental): Placebo group: The patient received the same dose of brown sugar water for 7 days before surgery. Folic acid dose selection is based on the maximum daily intake of children（tolerable upper intake levels，UL）
  Interventions: Drug: Folic Acid; Drug: Placebos

INTERVENTIONS:
Drug: Folic Acid — The patient was continuously taking 7 ml of a brown sugar aqueous solution containing a certain amount of folic acid for 7 days before surgery (0.3 mg/d for children with 1-3 years old and 0.4 mg/d for children aged 4 to 5, once a day). After the operation, the PAED scores were performed every 10 minutes during the recovery of the child, at the time of extubation, and within 30 minutes after extubation. The PAED scores of all the children were performed by the same measurer. (The total score is 0~20 points, and the score ≥10 points is defined as the recovery period).
Drug: Placebos — Patients in the placebo group received 20 ml of an aqueous solution of brown sugar with the same concentration as the intervention group on the 7th day before surgery. After the operation, the PAED scores were performed every 10 minutes during the recovery of the child, at the time of extubation, and within 30 minutes after extubation. The PAED scores of all the children were performed by the same measurer. (The total score is 0~20 points, and the score ≥10 points is defined as the recovery period).
  Arms: Placebo group

SUMMARY:
Research purposes：Comparison of preoperative folic acid and placebo intervention on postoperative recovery of sputum in children undergoing general anesthesia for head and neck and maxillofacial surgery Test type：Randomized, double-blind, placebo-controlled, prospective study Randomized grouping: Patients were randomized into an intervention group (fed for 7 days before surgery) and a placebo group (7 days for placebo) Test subjects: recruitment and sample size calculation, inclusion criteria, exclusion criteria, shedding cases, trial suspension, rejection criteria, trial termination,Test contents Evaluation indicators: main observation indicators, secondary observation indicators Adverse events: definition of adverse events, recording of adverse events, treatment of adverse events, assessment of adverse events, serious adverse events, definition of serious adverse events, recording and reporting of serious adverse events

DETAILED DESCRIPTION:
According to literature review, the incidence of sputum sputum in children is about 38.8% (Reference 1), and the incidence of sputum sputum in the placebo group is 38%, assuming a class of error probability α = 0.05, test efficiency 1-β=0.8, considering folic acid supplementation for 7 days can reduce the incidence of sputum to 23%. A chi-square test is proposed to assess whether there is a difference in the incidence of sputum between groups. Calculated by PASS software, the sample size was 300. Considering the 5% drop rate, a total of 316 inpatients with head and neck and maxillofacial surgery were included, divided into 2 groups, 158 cases in each group.

The PAED score was scored every 10 minutes during the recovery of the child, at the time of extubation, and within 30 minutes after extubation (total score 0-20, score ≥10 is defined as the recovery period).

8.2 secondary observation indicators:

1. Changes in induction of anesthesia, intubation, and central rate (HR) and mean blood pressure (MBP);
2. HR and MBP changes in the resuscitation chamber (T1), 5 min (T2) before extubation, T3 at extubation, and 2 min (T4) after extubation;
3. extubation time and wake-up time;
4. Postoperative Ramsay sedation scores were performed every 10 minutes during recovery, at the time of extubation, and within 30 minutes after extubation;
5. Postoperative pain CHEOPs scores were taken every 10 minutes during extubation and 30 min after extubation (the total score was less than 6 points and no pain was observed, and ≥10 points were treated with corresponding analgesia);
6. The use of anesthetic drugs (eg, pentazocine, propofol);
7. Changes of serum IL-6, TNF-α and folic acid concentrations before and after surgery.
8. Other adverse events during the recovery period (eg nausea and vomiting, bronchospasm, respiratory depression, etc.)

ELIGIBILITY:
Inclusion Criteria:

1. ASA is graded from I to II
2. Children between the ages of 1 and 5
3. The weight is greater than or equal to 8.5kg
4. It is planned to undergo head and neck and maxillofacial surgery under general anesthesia

Exclusion Criteria:

1. Children with a history of respiratory infection within 1 week
2. Children with congenital malformations such as congenital heart disease
3. Children with central nervous system diseases or those with mental disorders or mental disorders
4. Children with long-term use of sedative or analgesic drugs
5. Children with severe liver and kidney dysfunction
6. receiving folic acid supplementation therapy or taking related derivatives
7. Taking drugs that affect absorption in the past 1 month, such as sulfonamides, aspirin, etc.
8. Participated in other related clinical studies in the past 3 months

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2019-12-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of sputum in children | 8 days
  The incidence of sputum in children with major indicators was tested by chi-square test or exact probability method.

CONTACTS AND LOCATIONS:
Overall Officials: ren zhou, Doctor, Principal Investigator — shanghai Ninth People Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210